CLINICAL TRIAL: NCT06347952
Title: Mapping Arterial Perforators of the Nipple Areolar Complex and the Horizontal Septum During Mammoplasty
Brief Title: Mapping Arterial Perforators Within the Breast During Mammoplasty
Acronym: Map-total
Status: Completed | Type: Observational
Sponsor: Royal Marsden NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: SE1188
Record Dates: First submitted 2024-03-29; First posted 2024-04-04 (Actual); Last update posted 2024-04-04 (Actual); Status verified 2024-03

CONDITIONS: Breast Cancer
Keywords: oncoplastic surgery; therapeutic mammoplasty; breast reduction for cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Use of Acoustic and color imaging doppler during surgery for breast cancer — The intervention (post pilot study) is to systematically record the effect of routine use of acoustic as well as color imaging doppler during mammoplasty for breast cancer (for both the therapeutic and symmetrising breast reduction).

SUMMARY:
Breast cancer surgery can often be carried out as part of a breast reduction procedure known as 'therapeutic mammoplasty'. Where a woman has a breast with adequate volume, even larger cancers can be removed in an aesthetically acceptable way with re-shaping of the breast (often reduction and lift) incorporated into the cancer removal. An expectation and desire for most women is that the nipple and areola (known as the 'nipple-areolar complex' or NAC) is not only preserved, but re-positioned (usually lifted) to re-balance the overall aesthetic result.

In moving the NAC, the surgeon must ensure an adequate blood supply is maintained to preserve nourishment of the NAC tissue otherwise it can die (necrose) resulting in its removal. The tissue carrying the blood supply is known as a 'pedicle' and is fashioned by the surgeon for each patient during surgery.

We know as surgeons, that in most areas of anatomy of the human body there are variations in the pattern of blood vessels. The NAC blood supply is no exception. Yet for each individual patient, the only way to safely know these anatomical patterns is to map them before or during surgery.

A surgical tool utilising an aspect of ultrasound (known as doppler) is often used to locate visually (or by hearing) blood flow from blood vessels in operations where such knowledge is critical to the success of the procedure (for example DIEP-based breast reconstruction or chest wall perforator flaps).

We would like to evaluate the effectiveness of the routine use of doppler for NAC preservation during mammoplasty procedures to see if it gives the consultant surgeon and/or trainee a greater degree of confidence when shaping the NAC pedicle to preserve its blood supply.

In addition, we evaluate the training potential of patients undergoing symmetrising breast reduction, whereby the tissue removed is first mapped using acoustic doppler as for the NAC above.

DETAILED DESCRIPTION:
Despite breast cancer being one of the most frequent affecting women worldwide, it is also one of the most curable. Its multimodality treatment is based on surgery, radiotherapy and systemic therapy.

Breast conservation has evolved thanks to the utilization of mammoplasty techniques to achieve better aesthetic results - known collectively as 'oncoplastic' when applied to cancer surgery.

The key considerations in oncoplastic surgery are: tumour characteristics (extent, location) and reconstituting the aesthetically acceptable breast shape as well as nipple-areola complex (NAC) preservation. The former is vital to achieve clear resection margins to optimise local control. Planning is aided by imaging with ultrasound, mammography and often MRI. NAC preservation is a priority and expectation of patients and surgeons alike developed in the field of aesthetic breast surgery by plastic surgeons.

The attachment of any structure to the body by its nourishing blood supply (arteries and veins) is known as a 'pedicle'. The anatomy of the pedicle and its preservation is key to preservation of the NAC which has a well understood blood supply albeit with variations across patients and well-described patterns (ref). To preserve the NAC as part of a cancer resection and aesthetic breast re-shaping, a pedicle must be fashioned and the NAC successfully re-positioned to restore the aesthetic balance of the newly shaped (and often lifted) breast.

The aim of this study is to determine if by use of doppler (acoustic or colour flow modalities) to map the blood vessels supplying the NAC (for each individual patient), surgeons and trainees can construct a safe pedicle with greater confidence and ease, reducing the concern about diminishing its blood supply which could lead to NAC necrosis and loss. We would like to study the nipple blood supply as it pertains to each patient before surgery using acoustic doppler (AD) and colour doppler imaging (CDI). Each modality has its strengths and weaknesses and this evaluation aims to assess the contribution of each.

The most challenging part of therapeutic mammoplasty is the pre-operative planning. The surgeon must consider (1) localization of the tumour location and extent, (2) re-shaping of the remaining breast parenchyma and (3) placement of the vascularized the NAC and pedicle.

Several studies have been done regarding NAC vascularization and its variation between not only each person, but also each side (right versus left). Most studies were on cadavers3, MRI 4or CT angiography5. On the other hand, Seitz et al6 pointed out the predominancy of the NAC vascularization based on preoperative MRI in the breast without cancer. Specifically, they split all 56 breasts into 5 categories: type I medial, type II lateral, type III central, type IV inferior, and type V mixed. Moreover, they highlighted that the majority of NACs were supplied mostly by medial vessels. Basaran et al7 evaluated sixteen patients with severe gigantomastia and they marked the vessel locations before surgery by using Doppler ultrasonography.

Given the variation between people and their breasts, in this SE we would like to map preoperatively the NAC vascularization to understand if it could assist the surgeon's plan or even enable them to modify the NAC pedicle design. The mapping will be done by both CDI and AC. We will use both techniques to understand if there will be any difference in their accuracy and to determine if 1 modality alone will suffice.

Whilst both methods (acoustic and colour flow doppler) are used selectively in cases by some surgeons, this SE will specifically if routine use incorporated into the procedure will systematically facilitate pedicle design. The doppler carries no risk to the patient and is considered a tool to facilitate surgery rather than an intervention beyond standard of care.

Specifically, acoustic doppler (AC) - is a hand-held device, easy to use intra-operatively which gives an audible signal in real-time to enable marking of the exact location of a blood vessel at a given point (or along a specified line) within the tissue / under the skin.

Colour doppler imaging (CDI) will additionally give visual information which includes the calibre and depth of the vessel and enables the entire course of the vessel and any connections to be mapped relatively easily.

In reality, when the design and shaping of the NAC pedicle is undertaken during the operation, ideal placement / movement of this structure may be restricted by the surrounding tissue attachments which the surgeon may be fearful of dividing in case a critical artery is divided in the process (compromising the NAC perfusion). Knowing the exact location of the artery will give the surgeon confidence in knowing how far such tissue mobilisation can be safely undertaken.

Some therapeutic mammoplasties also involve creation of a 'secondary pedicle' which consists of breast tissue - again mobilised on a pedicle which must be moved within the breast to fill a defect created by the cancer resection. A secondary aim of this SE will be to map the principle arteries which supply that tissue as well.

In summary, this SE aims to establish the benefits of an ad-hoc practice by careful documentation of consecutive cases prospectively during surgery for mammoplasty where NAC or secondary pedicle mobilisation is required.

ELIGIBILITY:
Inclusion Criteria:

* female patients >18 years age
* plan for construction of at least 1 (i.e. unilateral / bilateral) NAC pedicle based on the superficial branches of either the 2nd (superior), 3rd (medial) anterior intercostal, the lateral thoracic (lateral) arteries or a combination thereof.

Exclusion Criteria:

* Patients planned solely for inferior NAC pedicle reduction mammoplasty
* patients planned for bilateral nipple/NAC sacrifice

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A prospective single-centre cohort study on consecutive patients diagnosed with primary breast cancer undergoing either therapeutic or symmetrising mammoplasty (Wise or vertical scar pattern) or both. Inclusion criteria were female patients >18 years age and plan for construction of at least 1 (i.e. unilateral / bilateral) NAC pedicle based on the superficial branches of either the 2nd (superior), 3rd (medial) anterior intercostal, the lateral thoracic (lateral) arteries or a combination thereof.
Sampling Method: Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2022-04-27 (Actual); Primary Completion 2024-01-25 (Actual); Study Completion 2024-01-29 (Actual)

PRIMARY OUTCOMES:
Full-thickness (complete or partial) necrosis of nipple-areolar complex | Within 30 days after surgery
  Any amount (as witnessed clinically) of full-thickness necrosis of the nipple-areolar complex of either breast in patients who have undergone breast reduction (for cancer - on the cancer side or matching reduction side)

CONTACTS AND LOCATIONS:
Overall Officials: Peter A Barry, MPhil, FRACS, Principal Investigator — Royal Marsden NHS Foundation Trust
Locations (1):
- Royal Marsden - Surrey, Sutton, England, United Kingdom